CLINICAL TRIAL: NCT06074510
Title: A Phase 4 Open-Label Multicenter Study of PYLARIFY® PET/CT or PET/MRI in Men With Newly Diagnosed Favorable Intermediate Risk (FIR) Prostate Cancer
Brief Title: PYLARIFY® PET/CT or PET/MRI in Men With Favorable Intermediate Risk (FIR) Prostate Cancer
Acronym: MIRROR
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PYL4301
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Favorable Intermediate Risk; PYLARIFY; PET
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PYLARIFY PET (Experimental)
  Interventions: Drug: Piflufolastat F 18 Intravenous Solution [PYLARIFY]

INTERVENTIONS:
Drug: Piflufolastat F 18 Intravenous Solution [PYLARIFY] — Participants will receive a single dose of 333 MBq (9 mCi) [296 MBq-370 MBq (8 mCi - 10 mCi)] PYLARIFY injection followed by a single whole-body PET/CT or PET/MRI scan acquired at 1 to 2 hours post-dosing
  Other Names: PYLARIFY; 18F-DCFPyL

SUMMARY:
The purpose of this study is to learn whether PYLARIFY PET imaging (study scan) can safely and accurately detect the presence or absence of prostate cancer growing beyond the prostate gland in men with favorable intermediate risk prostate cancer.

Participants will receive a single dose of PYLARIFY injection followed by a single whole-body PET/CT or PET/MRI scan acquired at 1 to 2 hours after PYLARIFY injection. Participants with positive study scan results that are suspicious for prostate cancer outside of the prostate gland may be asked to undergo additional diagnostic test(s) and/or recommend certain treatment(s) for prostate cancer within 2 to 90 days after the study scan. Participants will be monitored for up to 12 months to collecting information about treatment they receive for prostate cancer and results of regular PSA blood draws if ordered by doctors for up to 12 months after the study scan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and sign an approved informed consent form (ICF)
2. Patients must have the ability to understand and comply with all protocol requirements
3. Patients must be ≥ 18 years of age
4. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
5. Patients with life expectancy of at least 13 months as determined by the investigator
6. Patients must have confirmed favorable intermediate risk (FIR) adenocarcinoma of the prostate per 2023 NCCN guidelines. FIR risk group confirmation includes all the following:

   * 1 intermediate risk factor (cT2b-cT2c or ISUP Grade Group 2 or PSA 10-20 ng/mL)
   * ISUP Grade Group 1 or 2
   * <50% biopsy cores positive (e.g., <6 of 12 cores)

Note: Date of the prostate biopsy should be no sooner that 2 weeks and no later than 3 months prior to PYLARIFY PET imaging

Exclusion Criteria:

1. Patients administered any high energy (>300 KeV) gamma-emitting radioisotope within 5 physical half-lives prior to Day 1 (PYLARIFY imaging)
2. Previous Prostate cancer treatment including radiation, androgen deprivation therapy, brachytherapy, surgery, prostate ablation, hormonal therapies or investigational therapy
3. Known hypersensitivity to the components of PYLARIFY or its analogs
4. Patients with any medical condition or other circumstances that, in the opinion of the investigator, compromise the safety or compliance of the subject to produce reliable data or complete the study
5. Patients who have any radiographic evidence of T3, N1 or M1 disease on SOC imaging (if performed)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Detection rate | Day 1
  The proportion of participants with prostate cancer in whom PYLARIFY PET detected previously occult intraprostatic ISUP grade ≥3 lesions as assessed by pathology, or in whom PYLARIFY PET detected the presence of either/or extraprostatic extension, seminal vesicle invasion, regional lymph node involvement, distant metastases, divided by the number of subjects who undergo a PYLARIFY PET scan

SECONDARY OUTCOMES:
Change in intended patient clinical management | Day 30
  Intended medical management plan before and after PYLARIFY PET imaging
True detection rate | Day 1
  The percentage of participants with at least one true positive lesion identified on PYLARIFY PET imaging and confirmed by the truth standard. This measure includes patients in whom PYLARIFY PET detected previously occult intraprostatic ISUP grade ≥3 lesions as confirmed by pathology; or patients in whom PYLARIFY PET detected the presence of either/or extraprostatic extension, seminal vesicle invasion, regional lymph node involvement, distant metastases as assessed by central readers and verified by the standard of truth.
Correct localization rate | up to day 90
  The percentage of participants for whom there is a one-to-one correspondence on the same side between the location of at least one lesion outside of prostate capsule (extraprostatic extension, seminal vesicle invasion, pelvic lymph nodes, extrapelvic lymph nodes, extrapelvic bone or extrapelvic soft tissue lesion(s) identified on PYLARIFY PET/CT or PET/MR and the standard of truth.
Positive predictive value of PYLARIFY | up to day 90
  The percentage of participants who undergo PYLARIFY PET imaging that identifies a lesion or lesions outside of the prostate capsule and have an established standard of truth. Positive predictive value does not require a one-to-one correspondence by lesion location but requires that the lesion and standard of truth be within the same anatomic region, including prostatic, pelvic, extra-pelvic or distant lesions.
Sensitivity of PYLARIFY | up to day 90
  Sensitivity at the patient level for patients who undergo prostate surgery for prostate and with pelvic lymph nodes removal.
Specificity of PYLARIFY | up to day 90
  Specificity at the patient level for patients who undergo prostate surgery for prostate and with pelvic lymph nodes removal.
Negative predictive value of PYLARIFY | up to day 90
  Negative predictive value at the patient level for patients who undergo prostate surgery for prostate and with pelvic lymph nodes removal.
Number of participants with Adverse Events | Day 1

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Hoag Cancer Center, Irvine, California
  - Tower Urology, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - University of Iowa Health Care, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute Wayne State University, Detroit, Michigan
  - BAMF Health, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Huntsman Cancer Institute University of Utah, Salt Lake City, Utah